CLINICAL TRIAL: NCT05330182
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study of LMN-201 for Prevention of C. Difficile Infection Recurrence
Brief Title: LMN-201 for Prevention of C. Difficile Infection Recurrence
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lumen Bioscience, Inc. (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDI02; CDMRP-PR221885 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Clostridioides Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An open label sentinel cohort will be followed by a double-blind placebo-controlled main cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sentinel Cohort (Experimental)
  Interventions: Drug: LMN-201
- LMN-201 (Active Comparator)
  Interventions: Drug: LMN-201
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LMN-201 — LMN-201 consists of orally delivered whole, dried, non-viable biomass of spirulina (Arthrospira platensis) grown from 4 separate strains, each of which has been engineered to express one of the following therapeutic proteins:
  * 3 toxin-binding proteins that bind and inhibit C. difficile toxin B (TcdB), an essential virulence factor for C. difficile
  * 1 lysozyme-like enzyme that selectively degrades the cell wall of C. difficile and causes rapid destruction of the organism
  Arms: LMN-201; Sentinel Cohort
Drug: Placebo — Doses of placebo will be delivered as identical-appearing cornstarch with coloring in size 00, white, opaque, capsules.
  Arms: Placebo

SUMMARY:
This is a multisite study to evaluate the safety, tolerability, and efficacy of LMN-201 in participants recently diagnosed with CDI who are scheduled to receive or are receiving SOC antibiotic therapy against C. difficile.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 or older.
2. Diagnosis of CDI defined as a new or recent history of 3 or more bowel movements per day with a loose or watery consistency (Bristol Stool Scale 5, 6, or 7); a positive stool C. difficile toxin B immunoassay (stool collected no more than 7 days before first dose of LMN-201/placebo), and no other likely explanation for diarrhea. NOTE: Diarrhea is not required to be present on the day of enrollment.
3. Provision of signed and dated informed consent form.
4. Scheduled to receive or planning to receive a ≤28-day course of SOC antibiotic therapy for CDI. Participant must have been diagnosed with CDI for 7 or fewer days at time of initial study drug administration. SOC antibiotic therapy is defined as the receipt of oral fidaxomicin or oral metronidazole or oral vancomycin (see Section 8.2.6)
5. May be on systemic antibiotics for an infection unrelated to the gastrointestinal tract.
6. Ability to take oral medication and willingness to adhere to the study medication regimen.
7. Stated willingness and ability to comply with all study procedures and availability for the duration of the study and investigator believes individual will complete the study.
8. Access to a mobile smartphone.
9. For females of reproductive potential: use of highly effective contraception for at least 4 weeks prior to screening and agreement to use such a method during study participation and for an additional 4 weeks after the end of study drug administration.
10. For males of reproductive potential: agreement to use condoms or other methods to ensure effective contraception with partner during study participation and for an additional 4 weeks after the end of study drug administration.

Exclusion Criteria:

1. Fulminant C. difficile colitis.
2. Admitted or expect to be admitted to an intensive care unit.
3. Underlying gastrointestinal disorder characterized by diarrhea including but not limited to chronic ulcerative colitis, Crohn's disease, celiac sprue, short bowel syndrome, dumping syndrome following gastrectomy, pancreatic insufficiency, enteric parasitic infection, viral enteritis, bacterial enteritis (salmonella, shigella, ETEC, etc.).
4. Neutropenia (absolute neutrophil count of < 1000 per microliter for any reason).
5. Current or previous treatment in past 3 months with any therapy likely to influence the outcome of this study, including but not limited to the following:

   1. Bezlotoxumab (Zinplava, Merck & Co.), or another antibody against C. difficile toxin(s)
   2. C. difficile vaccine
   3. SER-109 (Seres Therapeutics)
   4. CP101 (Finch Therapeutics)
   5. VE303 (Vedanta Therapeutics)
   6. Fecal microbiota transplant
   7. Current therapy with oral exchange resins
   8. Protracted exposure to mu-agonist opioids and/or anticholinergic medication prescribed for diarrheal symptoms (unable to stop mu-agonist opioid treatment unless on a stable dose as of onset of diarrhea and no increase in dose planned for the duration of the study.)
6. Treatment with SOC antibiotic therapy is planned for longer than a 28-day period.
7. Pregnancy, anticipated pregnancy, or breastfeeding.
8. Inability or unwillingness to swallow numerous, relatively large capsules containing study drug or placebo because of a swallowing disorder or dysphagia.
9. Inability to pass swallowed capsules into the distal small intestine because of gastroparesis, repetitive vomiting, or anatomic narrowing in the esophagus, stomach, or small intestine.
10. Psychiatric illness that would affect compliance with medications, study capsules, or follow-up.
11. Status as an inmate, residential mental health program, or residential substance abuse program.
12. Terminal illness with limited life expectancy of less than 24 weeks.
13. Poor concurrent medical risks with clinically significant co-morbid disease such that, in the opinion of the investigator, the patient should not be enrolled.
14. Any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of the individual, would make it unlikely for the individual to complete the study, or would confound the results of the study.

    * Note: Use of probiotics and other food supplements (e.g., yogurt, kefir, kimchi, etc.) are not exclusionary.
    * Note: Assuming participants meet all of the inclusion criteria and none of the exclusion criteria, participants with underlying malignancy with a good life expectancy in the study are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve global cure | Up to 16 weeks after initiation of therapy
  Proportion of total participants with both successful initial CDI treatment and no CDI recurrence during the Prevention and Observation Phases (by treatment assignment).

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Kaiser Permanente, Escondido, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Gastroenterology Center of Connecticut, Hamden, Connecticut
  - GI PROS Research, Naples, Florida
  - Metro Infectious Disease Consultants - Atlanta, Decatur, Georgia
  - Snake River Research, Idaho Falls, Idaho
  - Metro Infectious Disease Consultants, LLC, Burr Ridge, Illinois
  - DM Clinical Research, Oak Lawn, Illinois
  - Baptist Health Research, Lexington, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - Mercury Street Medical, Butte, Montana
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Weill Cornell Medicine, New York, New York
  - IMA Clinical Research, Mount Airy, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Clinical Alliance for Infectious Diseases - Infectious Diseases, LLC, Annandale, Virginia

IPD SHARING:
Plan to Share IPD: No